CLINICAL TRIAL: NCT02247999
Title: Improving Cervical Cancer Prevention Among HIV-Infected Women Using Novel HPV Based Biomarker Assays
Brief Title: Improving Cervical Cancer Screening Among HIV-Infected Women in India
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913037; 13-C-N037
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Cervical Cancer; HIV/AIDS; HPV; Cervical Intraepithelial Neoplasia; Biomarkers
Keywords: Cervical Cancer; HIV/AIDS; HPV; Biomarkers; Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Cohort: HIV-infected women attending HIV care and treatment clinics in Pune, Chennai, andBelgaum in India.

SUMMARY:
Background:

* Cervical cancer is a major cause of cancer deaths among women. Most cases of cervical cancer are caused by the human papillomavirus (HPV). HPV is more common in women who have the human immunodeficiency virus (HIV). India has one of the highest rates of women who have both cervical cancer and HIV infection.
* Cervical cancer can be discovered in early stages by screening for HPV infection. Researchers want to compare new cervical cancer screening tests for HIV-infected women. They also want to know more about how HPV can lead to cervical cancer in HIV-infected women. To do so, they will hold a study to screen HIV-infected women in India.

Objectives:

- To improve cervical cancer screening methods in HIV-infected women in India.

Eligibility:

* Women at least 18 years of age who have HIV infection.
* Participants will be recruited from HIV-focused health care clinics in Pune and Chennai, India.

Design:

* Participants will have a physical exam and medical history. They will provide a urine sample and proof of HIV infection.
* Participants will have a gynecological exam. This will involve a pelvic exam and Pap smear to collect cells for study. It will also involve a cervical exam to look for precancerous cells. Cervical tissue may be collected.
* Participants will also provide a blood sample for testing.
* Participants will return in 2 weeks for the test results. If there are signs of precancerous or cancer cells, participants will be referred to a doctor for treatment.

DETAILED DESCRIPTION:
Background:

While HPV DNA testing is a highly sensitive screening method for cervical cancer, it cannot differentiate between the majority of benign infections and few persistent infections linked to cervical precancer. Given the high prevalence of carcinogenic HPV DNA and higher risk for cervical precancer and cancer among HIV-infected women, there is a substantial need for screening tests that are both adequately sensitive as well as specific, so as to maximize detection while reducing false-positive referrals. Furthermore, the unique immunological milieu in HIV-infected women presents significant opportunities to study natural history of HPV-mediated cervical oncogenic process in the context of immunosuppression.

Objectives and Methods:

The primary objective is to evaluate the clinical performance of two novel biomarker assays for detection of histologically-confirmed cervical intraepithelial neoplasia grade 2/3 or more severe (greater than or equal to CIN2 and greater than or equal to CIN3) among HIV-infected women. These tests include: (i) immunocytostaining by p16(INK4a)/Ki-67 (biomarkers correlated with the oncogenic transformation of cervical cells following persistent carcinogenic HPV infection) and (ii) testing for HPV E6/E7 mRNA (expressed during progression of a transient to a transforming HPV infection). Secondary objectives include studying the association of risk factors and biomarkers with specific HPV genotypes and studying the interaction of HIV and HPV in cervical disease categories and in the context of immunosuppression.

Eligibility:

HIV-infected women, 18 years or older, with no history of previous treatment for cervical precancer/cancer, not currently pregnant, and able to provide informed consent.

Design:

This cross sectional study will be conducted in collaboration with Indian Council of Medical Research (ICMR), in three institutions, with substantial experience in conduct of clinical research on HIV/AIDS and HPV/cervical cancer: the National AIDS Research Institute (NARI) in Pune, the National Institute of Epidemiology (NIE) in Chennai, and the Jawaharlal Nehru Medical College (JNMC) in Belgaum. A total of 1000 HIV-infected women attending HIV care and treatment clinics in Pune (n=400) and Chennai (n=400), and Belgaum (n=200) will be recruited. According to routine practice, participants will undergo per-speculum examination and cervical specimen collection, followed by a detailed diagnostic colposcopy exam with biopsies as indicated for histological analysis. Cervical specimens will be used for liquid-based cytology as well as simultaneous independent assessment with p16(INK4a)/Ki-67 and HPV E6/E7 mRNA testing. HPV DNA genotyping will be conducted by Linear Array HPV polymerase chain reaction. We will estimate the clinical performance (sensitivity, specificity, positive and negative predictive values, Youden s Index, and positive and negative likelihood ratios with 95% confidence intervals) of individual tests and combinations for prevalent detection of histologically-confirmed greater than or equal to CIN2 and greater than or equal to CIN3 among HIV-infected women. Additionally we will estimate age-specific and disease-specific HPV prevalence rates and HPV genotype composition, examine factors associated with greater than or equal to CIN2/greater than or equal to CIN3 lesions, examine the relationships of biomarker positivity at the HPV genotype-specific level, and evaluate the role of immunosuppression on HPV-mediated carcinogenesis. This study will permit validation of collection, transport, storage, and implementation protocols, allow evaluation of the field adoption and efficacy of these newer assays, describe the sensitivity and specificity of any of the tests or combinations with reasonable precision for a wide range of prevalence of greater than or equal to CIN3, and provide a resource for studies of HIV-HPV coinfection.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Female greater than or equal to 18 years of age at study entry. This ensures that all participants are at or above legal age in India for giving informed consent.
  2. Confirmed HIV-1 infection.
  3. For women of reproductive potential, a negative urine pregnancy test with a sensitivity of <25mlU/mL prior to study entry. This ensures that only non-pregnant women are included. While pregnancy is not an absolute contraindication for screening, certain invasive clinical procedures are often postponed until after pregnancy.
  4. If recently given birth, must be at least 12 weeks postpartum.
  5. Physical and mental ability and willingness of participant to provide written informed consent.

EXCLUSION CRITERIA:

1. Current or prior history of cervical, vaginal, or vulvar cancer.
2. Prior treatment for cervical disease; including treatment by cervical cryotherapy, LEEP, cervical conization, total or partial hysterectomy, chemotherapy, or radiation therapy.
3. Prior cervical procedure in the past 6 months, including dilatation and curettage (D&C).
4. Serious illness requiring systemic treatment or hospitalization within 21 days prior to study entry.
5. Active drug or alcohol use or dependence or any other condition that, in the opinion of the site investigator, would interfere with the participant s ability to adhere to study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from HIV-infected women attending HIV care and treatment clinics in Pune, Chennai, and Belgaum in India.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Cervical Intraepithelial Neoplasia Grade II or more severe | At enrollment
  Cervical Intraepithelial Neoplasia Grade II or more severe

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institute of Epidemiology (NIE), Chennai, India

REFERENCES:
- [Background] Sahasrabuddhe VV, Luhn P, Wentzensen N. Human papillomavirus and cervical cancer: biomarkers for improved prevention efforts. Future Microbiol. 2011 Sep;6(9):1083-98. doi: 10.2217/fmb.11.87. PMID 21958146
- [Background] Wentzensen N, Fetterman B, Castle PE, Schiffman M, Wood SN, Stiemerling E, Tokugawa D, Bodelon C, Poitras N, Lorey T, Kinney W. p16/Ki-67 Dual Stain Cytology for Detection of Cervical Precancer in HPV-Positive Women. J Natl Cancer Inst. 2015 Sep 15;107(12):djv257. doi: 10.1093/jnci/djv257. Print 2015 Dec. PMID 26376685
- [Background] Mane A, Nirmalkar A, Risbud AR, Vermund SH, Mehendale SM, Sahasrabuddhe VV. HPV genotype distribution in cervical intraepithelial neoplasia among HIV-infected women in Pune, India. PLoS One. 2012;7(6):e38731. doi: 10.1371/journal.pone.0038731. Epub 2012 Jun 19. PMID 22723879